CLINICAL TRIAL: NCT03433950
Title: Clinical Characteristics of Parkinson's Disease Subjects With Severe Hypertension During Motor OFFs.
Acronym: CLIN-HTN-PD
Status: Suspended | Type: Observational
Why Stopped: COVID-19 Research Restrictions
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kathryn Anne Chung, Prinicpal Investigator, Oregon Health and Science University
Other Study IDs: 17490; VA IRB 4143 (Other: VA Portland Health System)
Record Dates: First submitted 2018-01-08; First posted 2018-02-15 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease; Hypertension; Antiparkinsonism Drugs Causing Adverse Effects in Therapeutic Use
Keywords: antiparkinson
MeSH Terms: conditions — Parkinson Disease; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fluctuator: Parkinson's subjects with rises in systolic blood pressure exceeding 50% of baseline during motor off periods to select for subjects with severe blood pressure fluctuations.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Observational

SUMMARY:
Current management of hypertension in PD motor fluctuators is flawed. The current practice often is to treat transient hypertensive spikes reported by patients or measured in clinics with anti-hypertensive medications. This may contribute to morbidity by worsening orthostatic hypotension and increasing fall risk. There is a scarcity of literature on this subject and there is no documentation of severe hypertension with rises in systolic blood pressure exceeding 50% of baseline occurring during motor "OFF". There are two studies that have demonstrated that blood pressure fluctuation can occur in motor fluctuators during the "OFF" state1,2. The study by Baratti et al measured blood pressure in 13 Parkinson's disease patients, 7 with motor fluctuations and 6 without fluctuations. In the fluctuators, the mean systolic/diastolic blood pressures were significantly higher than the non-fluctuators during the "OFF" state but not the "ON" state.

DETAILED DESCRIPTION:
This is an observational study. This study will only recruit Parkinson's subjects with rises in systolic blood pressure exceeding 50% of baseline during motor off periods to select for subjects with severe blood pressure fluctuations. The clinical characteristics, including but not limited to, the degree of change of the motor tapping score, during an "off" period of this group of subjects with severe hypertension. There is a screening visit, a at home monitoring period, and a one-time 4-8 hour study visit for subjects that satisfy the inclusion criteria. The screening visit will assess Parkinson's motor state and review the inclusion/exclusion criteria. The at home monitoring period will measure blood pressure twice a levodopa cycle for 5 cycles (for most subjects, this will be for two days and is dependent on the subject's clinical levodopa cycle). Measurements will occur pre-levodopa dose (the maximal "OFF" time), and half-way through the cycle (maximal "ON" time). The percentage of change will be calculated and those that have a systolic change of greater than or equal to 50% will proceed to the outpatient visit. The outpatient visit will measure blood pressure, pulse, Parkinson's motor symptoms, and plasma levodopa levels.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease fulfilling UK Brain Bank clinical criteria.
* Treatment with chronic levodopa (levodopa treatment for ≥ 3 years).
* Rise in "OFF" systolic blood pressure exceeding 50% of baseline "ON" systolic blood pressure as shown by at home monitoring.
* History of "wearing off" prior to 4 hours after the previous levodopa dose per patient report or chart documentation.

Exclusion Criteria:

* Daily beta-blocker therapy.
* Diabetes mellitus, autonomic neuropathy, or other condition known to alter autonomic functions.
* Significant cognitive impairment as measured by the Montreal Cognitive Assessment score of < 16

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease participants with motor fluctuations.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure Change | Change in systolic blood pressure from 08:30 am measurement to 11:00 am measurement.
  Blood pressure measurement taken at lowest "OFF" rating on the Unified Parkinson's Disease Rating Scale (UPDRS) and highest "ON" rating on the UPDRS.

SECONDARY OUTCOMES:
Diastolic Blood Pressure Change | Change in systolic blood pressure from 08:30 am measurement to 11:00 am measurement.
  Blood pressure measurement taken at lowest "OFF" rating on the Unified Parkinson's Disease Rating Scale (UPDRS) and highest "ON" rating on the UPDRS.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baratti M, Calzetti S. Fluctuation of arterial blood pressure during end-of-dose akinesia in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1984 Nov;47(11):1241-3. doi: 10.1136/jnnp.47.11.1241. PMID 6502182
- [Result] Chase TN, Mouradian MM, Engber TM. Motor response complications and the function of striatal efferent systems. Neurology. 1993 Dec;43(12 Suppl 6):S23-7. PMID 8264907
- [Result] Pursiainen V, Korpelainen JT, Haapaniemi TH, Sotaniemi KA, Myllyla VV. Blood pressure and heart rate in parkinsonian patients with and without wearing-off. Eur J Neurol. 2007 Apr;14(4):373-8. doi: 10.1111/j.1468-1331.2007.01672.x. PMID 17388983